CLINICAL TRIAL: NCT00240721
Title: A Randomized, Double-Blind, Multicenter, Placebo-Controlled 12-Week Study Of The Safety And Efficacy Of Two Doses Of Topiramate For The Treatment Of Acute Manic Or Mixed Episodes In Subjects With Bipolar I Disorder With An Optional Open-Label Extension
Brief Title: A Study of the Effectiveness and Safety of Topiramate in the Treatment of Patients With Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002248
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-11

CONDITIONS: Bipolar Disorders; Mood Disorders; Affective Disorders, Psychotic
Keywords: topiramate; bipolar disorders; mood disorders; manic state; depression; manic-depressive psychoses
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Affective Disorders, Psychotic; Mania; Depression | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness and safety of topiramate compared with placebo in the treatment of acute manic or mixed episodes in patients with Bipolar I Disorder.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to evaluate the effectiveness of two dose levels of topiramate (400 and 600 milligrams/day) compared with placebo in the treatment of acute manic or mixed episodes in patients with Bipolar I Disorder. The trial consists of 3 phases: a screening period; double-blind treatment for 12 weeks; and an optional open-label period of at least 6 months. Assessment of effectiveness include change from baseline to Day 21 for the Young Mania Rating Scale (YMRS) total score. Also included during the 12 week study are the Global Assessment Scale (GAS), Montgomery-Åsberg Depression Rating Scale (MADRS), Brief Psychiatric Rating Scale (BPRS), Clinical Global Impressions (CGI), and health-related quality of life measures at specified time intervals. Safety assessments include evaluation of adverse events, rate of withdrawal from the study due to adverse events, and vital signs (blood pressure and pulse) throughout the study, as well as changes in clinical laboratory tests (hematology, biochemistry, urinalysis), electrocardiograms (ECGs), and physical examinations at specified times. The study hypothesis is that the change from baseline in Young Mania Rating Scale (YMSR) total score at Day 21 will be significantly better for the topiramate groups than for the placebo group. Topiramate tablets (50 or 100 milligrams) or placebo, beginning at 50mg daily and increasing over the first week to a maximum of 400mg/day or 600mg/day, depending on study group. Maximum dosage continues up to 12 weeks. Dosage can be decreased or increased at investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar I Disorder by criteria of Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV), and currently experiencing a manic or mixed episode by DSM-IV and Structured Clinical Interview criteria
* experienced at least one previous manic or mixed episode
* Young Mania Rating Scale (YMSR) score >=20
* physically healthy
* females must be postmenopausal, surgically sterile, or using adequate contraceptive measures, and have a negative pregnancy test.

Exclusion Criteria:

* Diagnosis of alcohol or substance dependence (with the exception of nicotine or caffeine dependence) by DSM-IV criteria
* DSM-IV Axis I diagnosis of schizoaffective disorder or impulse control disorder
* experienced a manic episode while taking an antidepressant or psychostimulant drug
* no significant and untreated or unstable medical illness of the liver, kidney, heart, lungs, or endocrine system
* no hypersensitivity to topiramate or have previously participated in a topiramate study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2000-10; Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 21 for the Young Mania Rating Scale (YMRS) total score.

SECONDARY OUTCOMES:
Change from baseline to Day 21 for scores on MADRS, BPRS, CGI, and GAS; response to treatment, indicated by not any longer meeting DSM-IV criteria for manic/mixed episode.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the effectiveness and safety of topiramate in the treatment of patients with Bipolar Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=464&filename=CR002248_CSR.pdf